CLINICAL TRIAL: NCT01256541
Title: A Single Center, Open-Label, Pilot Study to Determine the Safety, Efficacy, and Patient Preference of Kristalose as a Bowel Evacuant Prior to Colonoscopy
Brief Title: Kristalose as Bowel Evacuant Prior to Colonoscopy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other); Cumberland Pharmaceuticals (Industry)
Responsible Party: Otto Lin, MD, Virginia Mason Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB10068
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Bowel Evacuant Prior to Colonoscopy
MeSH Terms: interventions — Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kristalose (Experimental): Kristalose as Bowel Evacuant
  Interventions: Drug: Kristalose

INTERVENTIONS:
Drug: Kristalose — The dosing regimen of Kristalose will be nine 20-gram doses (one dose every 30 minutes for 4 straight hours) taken the evening before the colonoscopy procedure.

SUMMARY:
To determine whether Kristalose causes a significant increase in hydrogen and/or methane gas levels in patients requiring bowel evacuation, and also to determine the safety, efficacy, and patient preference of Kristalose as a bowel evacuant

DETAILED DESCRIPTION:
This is a single center, open-label, pilot study to determine the safety, efficacy, and patient preference of Kristalose as a bowel evacuant prior to colonoscopy. Prior to colonoscopy, subjects will also undergo evaluation for the production of hydrogen and methane gases in the patient's gut (before and after receiving Kristalose) as assessed by a breath analysis instrument. Safety will be assessed by the occurrence of any treatment emergent adverse events. Efficacy will be determined by the endoscopist's rating of the cleanliness of the colon and the incidence of treatment failure (insufficient evacuation of the bowel).

ELIGIBILITY:
Inclusion Criteria:

Patients requiring bowel evacuation for colonoscopy

Exclusion Criteria:

1. Patients with galactosemia (galactose-sensitive diet).
2. Patients known to be hypersensitive to any of the components of Kristalose.
3. Patients with possible bowel obstruction, previous colonic surgery, gastric retention, bowel perforation, toxic colitis, toxic megacolon, or ileus.
4. Patients less than 18 years of age.
5. Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]) and agree to abide by the study restrictions.
6. Be pregnant or nursing
7. Be otherwise unsuitable for the study, in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Hydrogen and Methane Gas Production | 3 months
  To evaluate the primary objective of hydrogen and methane gas production as measured by:
  • Pre- and post-dose breath analysis for hydrogen and methane gas.

SECONDARY OUTCOMES:
Efficacy | 3 months
  To evaluate the secondary objective of efficacy, the following endpoints will be measured:
  * Physician's determination of the cleanliness of the colon will be evaluated by completion of the Boston bowel prep scale.[4]
  * The number and percentage of patient's who by the physician's determination are considered treatment failures (patients with insufficient evacuation of the bowel=Boston bowel prep score < 5, and/or any colon segment score of 0).

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States